CLINICAL TRIAL: NCT06216223
Title: Surgery Versus Laser Ablation of Anal Diseases in Inflammatory Bowel Disease Patients
Brief Title: Laser Versus Surgery in Anal Diseases in Inflammatory Bowel Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #101080-5-9-2023
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases; Anal Fissure; Hemorrhoids
Keywords: anal fissure; hemorrhoids; inflammatory bowel disease; crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Fissure in Ano; Hemorrhoids; Crohn Disease; Colitis, Ulcerative | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser (Active Comparator): laser ablation of anal diseases in inflammatory bowel patients
  Interventions: Procedure: treatment of anal diseases in inflammatory bowel patients; Device: Laser
- traditional surgery (Sham Comparator): traditional surgery for anal diseases in inflammatory bowel patients
  Interventions: Procedure: treatment of anal diseases in inflammatory bowel patients; Procedure: traditional surgery

INTERVENTIONS:
Procedure: treatment of anal diseases in inflammatory bowel patients — treatment of anal diseases in inflammatory bowel patients
Device: Laser — laser
  Arms: laser
Procedure: traditional surgery — traditional surgery
  Arms: traditional surgery

SUMMARY:
This is a randomized comparative clinical trial carried out to compare between laser ablation and surgery in treating anal diseases in inflammatory bowel diseases patients and find out if one is superior to the other.

Inflammatory bowel diseases patients with anal problems were divided into 2 groups, one group had traditional surgery and the other had laser ablation for anal diseases and results were compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of inflammatory bowel disease ( non specific colitis, crohn's disease, ulcerative colitis).
* Patients who accidently discovered to have inflammatory bowel disease.
* Age group between 18 to 60 years old

Exclusion Criteria:

* Informed consent refusal.
* Proved malignancy in inflammatory bowel disease patients
* Patients less than 18 years old or more than 60 years old
* Contraindications to general and spinal anesthesia
* other types of colitis as ischemic colitis, pseudo-membranous colitis, infective colitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Operation time | Intraoperative (from skin incision to wound dressing.)
  operation time in minutes was studied between the 2 groups
operative bleeding | Intraoperative to 2 weeks after operation.
  bleeding in cc was calculated between the 2 groups
post operative anal discharge | from incision to 2 weeks after operation.
  presence of post operative anal discharge was detected in the 2 groups
pain score with visual analogue scale | from the 1st day to 2 weeks postoperatively
  pain score with visual analogue scale was studied between the 2 groups,minimum score is 0 which means painless and maximum score is 10 which means very painful
Healing time | healing time was studies from the 1st day to 3 months after operation
  time for complete healing after operation was studied between the 2 groups
Return to work | Return to work was assessed from one day to 2 months after surgery
  Return to work after operation was studied between the 2 groups
patient satisfaction score | from one day to 3 months after operation
  patient satisfaction score among patients in the 2 groups was studied using customer satisfaction score, minimum score is 1 means very dissatisfied and maximum score is 10 means very satisfied
Recurrence | detection of recurrence from 3 to 6 months after operation
  recurrence between 2 groups was assessed
Fistula occurence | from 2 weeks to 2 months after operation
  fistula occurence studied between the 2 groups
Stenosis | stenosis was detected from wound healing to 6 months later
  post operative stenosis between the 2 groups was studied
Discharge from hospital | from one day post operative to one week
  hospital stay studied between the 2 groups

SECONDARY OUTCOMES:
age | age of participants was recorded for one year duration of the study
  age in the 2 groups was studied
sex | sex of participants was recorded for one year duration of the study
  sex was studied in the 2 groups
specific disease | diagnosis of diseases known 2 days before surgery from history
  diagnosis of crohn's disease, ulcerative colitis, non specific colitis by colonoscopy and biopsy was done in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Reham Zakaria, PhD, Principal Investigator — faculty of medicine Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

REFERENCES:
- [Derived] Zakaria R, Amin MM, Abo-Alella HA, Hegab YH. Laser hemorrhoidoplasty versus hemorrhoidectomy in the treatment of surgically indicated hemorrhoids in inflammatory bowel patients: a randomized comparative clinical study. Surg Endosc. 2025 Jan;39(1):249-258. doi: 10.1007/s00464-024-11351-3. Epub 2024 Nov 7. PMID 39511001